CLINICAL TRIAL: NCT05712707
Title: Phase 1B Study of Sublingual Dexmedetomidine, an Alpha 2 Adrenergic Agonist, for Treating Opioid Withdrawal
Brief Title: Sublingual Dexmedetomidine for Treating Opioid Withdrawal
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: BioXcel Therapeutics Inc (Industry); Yale University (Other); Clinilabs, Inc. (Other); National Institute on Drug Abuse (NIDA) (NIH); CenExel HRI (Unknown)
Responsible Party: Principal Investigator, Sandra D. Comer, Clinical Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8325; UG3DA056247-01 (NIH)
Record Dates: First submitted 2023-01-24; First posted 2023-02-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder; Opioid Withdrawal
MeSH Terms: conditions — Opioid-Related Disorders | interventions — lofexidine

STUDY DESIGN:
Intervention Model Description: Throughout the 7-day inpatient study, participants will receive sublingual BXCL501 or placebo twice daily and lofexidine or placebo 4 times daily using a double-blind, triple-dummy design. This study will utilize a methadone taper in order to ensure that opioid withdrawal severity is not so severe that it results in discharge immediately after enrollment (before a medication effect can be observed). Throughout the 7-day inpatient study, participants will receive: Methadone QID at 9am, 2pm, 7pm, 11pm. Total daily methadone doses: Day 1= 30mg, Day 2= 25mg, Day 3= 20mg, Day 4= 15 mg, Day 5= 10mg, Day 6= 5mg, Day 7= 0mg. On each day a PRN methadone dose of 5mg x 2, will also be available (total daily dose will not exceed 40mg).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The current study is a randomized, double-blind, double-dummy inpatient study comparing BXCL501 (180 and 240 ug BID), lofexidine (as a positive control), and placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BXCL501 (180 micrograms) (Experimental): The current study is a randomized, double-blind, double-dummy inpatient study comparing BXCL501 (180 and 240 ug BID), lofexidine (as a positive control), and placebo.
  Interventions: Drug: BXCL501 (180 micrograms)
- BXCL501 (240 micrograms) (Experimental): The current study is a randomized, double-blind, double-dummy inpatient study comparing BXCL501 (180 and 240 ug BID), lofexidine (as a positive control), and placebo.
  Interventions: Drug: BXCL501 (240 micrograms)
- Lofexidine (Positive Control) (Active Comparator): The current study is a randomized, double-blind, double-dummy inpatient study comparing BXCL501 (180 and 240 ug BID), lofexidine (as a positive control), and placebo.
  Interventions: Other: Lofexidine (Positive Control)
- Placebo (Placebo Comparator): The current study is a randomized, double-blind, double-dummy inpatient study comparing BXCL501 (180 and 240 ug BID), lofexidine (as a positive control), and placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BXCL501 (180 micrograms) — Throughout the 7-day inpatient study (Figure 1; Table 1), participants will receive sublingual BXCL501 or placebo twice daily and lofexidine or placebo 4 times daily using a double-blind, double-dummy design.
  Arms: BXCL501 (180 micrograms)
Drug: BXCL501 (240 micrograms) — Throughout the 7-day inpatient study (Figure 1; Table 1), participants will receive sublingual BXCL501 or placebo twice daily and lofexidine or placebo 4 times daily using a double-blind, double-dummy design.
  Arms: BXCL501 (240 micrograms)
Other: Placebo — Throughout the 7-day inpatient study (Figure 1; Table 1), participants will receive sublingual BXCL501 or placebo twice daily and lofexidine or placebo 4 times daily using a double-blind, double-dummy design.
  Arms: Placebo
Other: Lofexidine (Positive Control) — Throughout the 7-day inpatient study (Figure 1; Table 1), participants will receive sublingual BXCL501 or placebo twice daily and lofexidine or placebo 4 times daily using a double-blind, double-dummy design.
  Arms: Lofexidine (Positive Control)

SUMMARY:
A major challenge to seeking treatment for opioid use disorder (OUD) is the withdrawal symptoms associated with cessation of opioid use. The signs and symptoms of opioid withdrawal include irritability, anxiety, muscular and abdominal pains, chills, nausea, diarrhea, yawning, runny eyes and nose, sweating, sneezing, weakness, and insomnia. The current gold standard of treatment involves a gradual reduction of the opioid drug dosage (tapering). However, as all opioids have potential for abuse and require careful dosing due to side effects (e.g., respiratory depression), a non-opioid medication to facilitate withdrawal severity would be of great value. Commonly used non-opioid medications like lofexidine have concerning side effects including sedation and low blood pressure. BioXcel Therapeutics has developed BXCL501 (dexmedetomidine: sublingual film) to reduce symptoms associated with opioid withdrawal. Dexmedetomidine is currently used as an intravenous anesthetic for its anxiety-reducing, sedative, and analgesic properties. The current study will seek to compare the safety and efficacy of BXCL501 relative to lofexidine and placebo in subjects with OUD who are physically dependent on opioids. Throughout a 7-day inpatient withdrawal period (using a methadone taper) opioid-dependent participants will receive sublingual BXCL501, placebo, or lofexidine. In comparison to lofexidine, dexmedetomidine is expected to have a superior safety profile with limited adverse effects on blood pressure and heart rhythm. Three sites will participate in this study: NYSPI, Clinilabs, Inc., and Yale University.

The NYSPI site is currently paused and has been paused since an institutional pause on human subjects research began in June 2023. The U.S. Department of Health and Human Services (HHS) Office of Human Research Protections (OHRP) issued an FWA restriction on NYSPI research that also included a pause of human subjects research as of June 23, 2023.

DETAILED DESCRIPTION:
A major challenge to seeking treatment for OUD is the withdrawal syndrome associated with cessation of opioid use. Withdrawal symptoms include irritability, anxiety, muscular and abdominal pains, chills, nausea, diarrhea, yawning, lacrimation, sweating, sneezing, rhinorrhea, general weakness, and insomnia. The intensity of withdrawal symptoms is one of the most common barriers to entering and completing treatment for patients, particularly those who may be interested in maintenance therapy with naltrexone, an opioid antagonist, or buprenorphine, an opioid partial agonist. Because of the short half-life of most illicitly used opioid drugs, such as heroin, withdrawal symptoms reach peak intensity within two to four days after last use, and the duration of withdrawal symptoms usually lasts 7-12 days (Antoine et al., 2021; Cook, 2021).

Currently, there are 2 major strategies to treat withdrawal symptoms after stopping opioid use: Gradual tapering using an opioid drug substitute (methadone or buprenorphine) and amelioration of withdrawal symptoms using alpha-2-adrenergic agonists and other non-opioid medications (benzodiazepines, nonsteroidal anti-inflammatory drugs, etc.) The current gold standard involves gradual reduction of the opioid drug dosage (tapering). The most common opioid withdrawal method is substituting and tapering with methadone or buprenorphine (Srivastava et al., 2020). These are opioid medications with longer half-lives than street opioids and result in more manageable withdrawal symptoms after stopping their use. However, buprenorphine and methadone can be diverted for illicit use, and is associated with adverse events such as respiratory depression, which could be further aggravated by concomitant drug and alcohol use in this population. Furthermore, discontinuation of opioid medications can lead to withdrawal symptoms. A non-opioid medication to facilitate withdrawal suppression from opioid discontinuation in OUD would be of great value.

For over four decades, studies have demonstrated that norepinephrine regulates activity of locus coeruleus neurons, the same neurons that are affected by opioid drugs (Maze et al., 1988). In 1978, several groups reported early successful experience with the use of the alpha-2a-adrenergic agonist clonidine to treat symptoms of opioid withdrawal (Cedarbaum & Aghajanian, 1977; Gold et al., 1978), which has led to their widespread use for this indication. Opioid physical dependence and withdrawal are mediated at least in part by the interaction of mu-opioid receptors with neurons that contain the neurotransmitter norepinephrine.

Activation of mu-opioid receptors normally suppresses the release of norepinephrine from the locus coeruleus. When opioid use is discontinued or blocked, the locus coeruleus releases excess norepinephrine, and this excess norepinephrine causes many of the withdrawal symptoms noted above. By administering an alpha-2a-adrenergic agonists (like lofexidine, clonidine and dexmedetomidine), hyperactivity of locus coeruleus neurons can be blocked and withdrawal symptoms reduced.

Lofexidine is currently approved in the U.S. for the mitigation of withdrawal symptoms during discontinuation from use of opioids under the brand name Lucemyra. In a recent clinical trial of lofexidine, only 41.5% of the participants taking lofexidine and 27.8% of patients on placebo completed the trial (FDA Approval 2018; Fishman et al., 2019). As a result, patients seeking treatment for illicit opioid use only have an ~4 in 10 chance of completing treatment with the only currently available non-opioid medication, lofexidine. Dexmedetomidine possesses superior pharmacological properties within the alpha-2-adrenergic agonist class. Dexmedetomidine is a full agonist with higher affinity for alpha-2a-adrenergic receptors compared to lofexidine and may be expected to produce a higher level of efficacy (Peltonen et al., 1998, Ouchi & Sugiyama, 2016; Zhang et al., 2013). *BXCL501 (120 and 180 mcg: IgalmiTM) was recently FDA approved for the acute treatment of agitation associated with schizophrenia or bipolar I or II disorder in adults.*

Few direct comparisons have been made between dexmedetomidine and lofexidine, but a recent meta-analysis comparing peri-operative adverse events related to dexmedetomidine versus clonidine showed that hypotension was similar for the 2 medications pre- and post-operatively but dexmedetomidine appeared to be protective against hypertension and tachycardia during surgery (Demiri et al., 2019). Furthermore, a trial directly comparing dexmedetomidine (n=144) and clonidine (n=142) in older adults undergoing cardiac surgery showed that dexmedetomidine had superior outcomes with regard to risk and duration of delirium, duration of mechanical ventilation, length of stay in the intensive care unit, mortality rate, and morphine consumption (Shokri & Ali, 2019). In summary, sublingual dexmedetomidine (BXCL501) is expected to be superior safety and efficacy to other alpha-2a-adrenergic agonists in the treatment of opioid withdrawal.

This study will be first direct comparison of BXCL501 to lofexidine on these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and complying with the protocol.
* 18 years of age or older but less than 60 years old.
* Has opioid use disorder moderate-to-severe (304.00) as per DSM-V, and physiological dependence on opioids.
* Females agree to use an acceptable method of contraception for the duration of the study.

Exclusion Criteria:

* Positive urine or serum pregnancy test at screening, after admission, planning to become pregnant during the course of the trial, or currently breast feeding.
* Clinically significant history of cardiac disease, including syncope, bradycardia, conduction abnormalities, orthostatic hypotension or blood pressure disorders. Heart rate and blood pressure at screening and baseline of < 50 beats per minute or systolic blood pressure <105, >150 mmHg or diastolic BP <70, >90 mmHg.
* Clinically significant medical condition or observed abnormalities (including: physical examination, hypotension, laboratory evaluation, and/or urinalysis findings). Clinically significant abnormal ECG such as second- or third-degree heart block, uncontrolled arrhythmia, or QTc interval > 450 msec for males, and > 470 msec for females.
* Evidence of hepatic abnormalities, including: ascites, bilirubin >10% above upper limit of normal and/or esophageal variceal disease, active hepatitis/aspartate aminotransferase, alanine aminotransferase >3x the upper limit of normal.
* Any psychiatric disorder that would compromise ability to complete study requirements [e.g. severe acute depression, active mania, or suicidality with specific plan and intent (assessed using the CSSRS)].
* Not being able to provide a negative urine for methadone or buprenorphine at screening.
* Use of oral naltrexone for ≥7 consecutive days within 60 days prior to screening.
* Need for alcohol or benzodiazepine detoxification.
* Participation in a clinical trial of a pharmacological agent within 30 days prior to screening.
* Use of any concomitant medication at screening or anticipated/required use during the study period that the investigators feel may impact participant safety or interfere with the aims of the trial (e.g., daily licit or illicit benzodiazepine use).
* Any finding that, in the view of the principal investigator, would compromise the subject's ability to fulfill the protocol visit schedule or visit requirements.
* Investigator-site personnel or immediate family of investigator-site personnel.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety of BXCL501 versus Placebo and Lofexidine | Study Days 1-7
  Establish the safety of BXCL501 relative to placebo and lofexidine in subjects with OUD who are physically dependent on opioids as measured by the frequency of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Comer, Ph.D, Principal Investigator — Columbia University / New York State Psychiatric Institute
Locations (4):
- United States (4):
  - Yale University, New Haven, Connecticut
  - Clinilabs, Eatontown, New Jersey
  - CenExel HRI, Marlton, New Jersey
  - New York State Psychiatric Institute, New York, New York

REFERENCES:
- [Background] Antoine D, Huhn AS, Strain EC, Turner G, Jardot J, Hammond AS, Dunn KE. Method for Successfully Inducting Individuals Who Use Illicit Fentanyl Onto Buprenorphine/Naloxone. Am J Addict. 2021 Jan;30(1):83-87. doi: 10.1111/ajad.13069. Epub 2020 Jun 23. PMID 32572978
- [Background] Srivastava AB, Mariani JJ, Levin FR. New directions in the treatment of opioid withdrawal. Lancet. 2020 Jun 20;395(10241):1938-1948. doi: 10.1016/S0140-6736(20)30852-7. PMID 32563380
- [Background] Maze M, Segal IS, Bloor BC. Clonidine and other alpha2 adrenergic agonists: strategies for the rational use of these novel anesthetic agents. J Clin Anesth. 1988;1(2):146-57. doi: 10.1016/0952-8180(88)90034-7. PMID 2908485
- [Background] Cedarbaum JM, Aghajanian GK. Catecholamine receptors on locus coeruleus neurons: pharmacological characterization. Eur J Pharmacol. 1977 Aug 15;44(4):375-85. doi: 10.1016/0014-2999(77)90312-0. No abstract available. PMID 330174
- [Background] Fishman M, Tirado C, Alam D, Gullo K, Clinch T, Gorodetzky CW; CLEEN-SLATE Team. Safety and Efficacy of Lofexidine for Medically Managed Opioid Withdrawal: A Randomized Controlled Clinical Trial. J Addict Med. 2019 May/Jun;13(3):169-176. doi: 10.1097/ADM.0000000000000474. PMID 30531234
- [Background] Shokri H, Ali I. A randomized control trial comparing prophylactic dexmedetomidine versus clonidine on rates and duration of delirium in older adult patients undergoing coronary artery bypass grafting. J Clin Anesth. 2020 May;61:109622. doi: 10.1016/j.jclinane.2019.09.016. Epub 2019 Oct 23. PMID 31668468